CLINICAL TRIAL: NCT00097266
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Study of Aripiprazole Monotherapy in the Treatment of Acutely Manic Patients With Bipolar I Disorder
Brief Title: Study of Aripiprazole in Patients With Acute Bipolar Mania
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-162
Record Dates: First submitted 2004-11-19; First posted 2004-11-22 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2010-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Mania
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole; Haloperidol

ARMS (3):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Experimental)
  Interventions: Drug: Aripiprazole
- C (Active Comparator)
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Placebo — Tablets/capsules, oral, 0 mg, once daily, 3 weeks (switched to arm B for an additional 9 weeks).
  Arms: A
Drug: Aripiprazole — Tablets, oral, 15-30 mg, once daily, 12 weeks.
  Other Names: Abilify
  Arms: B
Drug: Haloperidol — Capsule, oral, 5-15 mg, once daily, 12 weeks.
  Arms: C

SUMMARY:
The purpose of this research study is to confirm the safety and effectiveness of aripiprazole therapy over 12 weeks in subjects with bipolar disorder experiencing symptoms of mania.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Bipolar I Disorder and a diagnosis of acute mania will be considered for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615
Dates: Start 2004-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change in a mania rating scale at endpoint

SECONDARY OUTCOMES:
Response rate and Clinical Global Impression scale at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (45):
- United States (15):
  - Local Institution, Anaheim, California
  - Local Institution, Cerritos, California
  - Local Institution, Garden Grove, California
  - Local Institution, National City, California
  - Local Institution, Pico Rivera, California
  - Local Institution, Riverside, California
  - Local Institution, San Diego, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Maitland, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Cleveland, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, DeSoto, Texas
- Bulgaria (5):
  - Local Institution, Burgas
  - Local Institution, Novi Iskar
  - Local Institution, Pleven
  - Local Institution, Sofia
  - Local Institution, Varna
- Croatia (4):
  - Local Institution, Osijek
  - Local Institution, Rijeka
  - Local Institution, Split
  - Local Institution, Zagreb
- Mexico (7):
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Col. Obispado, Nuevo León
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Fracc. Industrias, San Luis Potosí
  - Local Institution, Mérida, Yucatán
  - Local Institution, Nuevo León
- Local Institution, Lima, Lima Province, Peru
- Russia (9):
  - Local Institution, Lipetsk, Lipetsk Oblast
  - Local Institution, Arkhangelsk
  - Local Institution, Kazan'
  - Local Institution, Leningrad Region
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Volgograd
- South Africa (4):
  - Local Institution, Florida, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Berea, Kwa Zuluu Natal
  - Local Institution, Durban, KwaZulu-Natal

REFERENCES:
- [Background] Young AH, Oren DA, Lowy A, McQuade RD, Marcus RN, Carson WH, Spiller NH, Torbeyns AF, Sanchez R. Aripiprazole monotherapy in acute mania: 12-week randomised placebo- and haloperidol-controlled study. Br J Psychiatry. 2009 Jan;194(1):40-8. doi: 10.1192/bjp.bp.108.049965. PMID 19118324